CLINICAL TRIAL: NCT01503840
Title: Evaluation of Accelerometer-Based Neuromuscular Monitoring Reliability to Exclude Postoperative Residual Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Federico Piccioni, MD, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: INT-66/11
Record Dates: First submitted 2011-12-29; First posted 2012-01-04 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Postoperative Residual Paralysis
MeSH Terms: interventions — Sugammadex; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Sugammadex (Active Comparator)
  Interventions: Drug: sugammadex
- Sodium chloride solution (Placebo Comparator)
  Interventions: Drug: Sodium chloride solution

INTERVENTIONS:
Drug: sugammadex — sugammadex 10 mg/ml diluted solution dosage: 1mg/kg i.v. (0,1 ml/kg)
  Other Names: Bridion
  Arms: Sugammadex
Drug: Sodium chloride solution — Sodium chloride solution 0,9% dosage: 0,1 ml/kg i.v.
  Arms: Sodium chloride solution

SUMMARY:
Accelerometer-based neuromuscular monitoring is not the gold-standard method to evaluate residual postoperative paralysis but it represents the most simple, inexpensive and widespread tool in clinical practice. Train-of-four ratio (TOF-ratio) of 100% is considered the gold-standard to avoid PORC (post operative residual curarization).

This clinical trial is conducted to verify the reliability of accelerometer-based neuromuscular monitoring in order to exclude postoperative residual paralysis which is not highlighted by this instrument at a TOF-ratio=100%.

The study evaluates patients' neuromuscular recovery evaluated using pulmonary function tests after extubation at a TOFratio=100%. Administering placebo or sugammadex at a TOF ratio=100% allows to evaluate whether the recovery of muscle function is concrete, although the monitoring device shows a complete decurarization; patients treated with sugammadex should not be capable to perform better pulmonary function tests if a TOF ratio=100% is reliable.

DETAILED DESCRIPTION:
From the beginning of the surgery to the time of extubation neuromuscular block is monitored with accelerographic monitor TOF-Watch SX. Patients are extubated when TOF-ratio is 100%.

Patients will perform pulmonary function tests (PFTs):

* the day ahead of surgery (for elegibility and training)
* 60 minutes before surgery
* 10 minutes after extubation
* 5 minutes after sugammadex or placebo administration
* 20 minutes after sugammadex or placebo administration.

The following parameters will be evaluated and compared between the 2 groups:

* Maximal Inspiratory Pressure (MIP)
* Maximal Expiratory Pressure (MEP)
* Forced Expiratory Volume in the first Second (FEV1)
* Forced Vital Capacity (FVC)
* Ratio of Maximum Expiratory Flow and Maximum Inspiratory Flow rate at 50% of vital capacity (MEF50/MIF50)
* PaO2, PaCO2, pH
* heart rate, blood pressure and respiratory rate

Changes of pulmonary tests performed before and after sugammadex or placebo will be compared between study groups.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing major abdominal surgery
* age between 18 and 70 years
* ASA class 1 or 2
* patients scheduled for blended anesthesia (epidural + general anesthesia)
* patients capable to perform pulmonary function tests (preoperative values of MIP, MEP, FEV1% and FEV1/FVC in normal ranges).

Exclusion Criteria:

* known or suspected respiratory, cardiovascular or neuromuscular disease
* renal or hepatic failure
* known or suspected allergies to drugs used in the study
* risk for malignant hyperthermia
* pregnancy
* diagnosed depressive disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)
Maximum Expiratory Pressure (MEP) changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)
Forced Expiratory Volume after the first second (FEV1) changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)
Forced Vital Capacity (FVC) changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)

SECONDARY OUTCOMES:
Ratio of Maximum Expiratory Flow and Maximum Inspiratory Flow rate at 50% of vital capacity (MEF50/MIF50) changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)
Hemogasanalysis parameters changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)
Swallow ability changes after placebo or sugammadex | 10 minutes after surgery and 5 minutes later
  10 minutes after surgery and 5 minutes later (after placebo or sugammadex administration)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Piccioni, MD, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori - Milan
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Result] Piccioni F, Mariani L, Bogno L, Rivetti I, Tramontano GT, Carbonara M, Ammatuna M, Langer M. An acceleromyographic train-of-four ratio of 1.0 reliably excludes respiratory muscle weakness after major abdominal surgery: a randomized double-blind study. Can J Anaesth. 2014 Jul;61(7):641-9. doi: 10.1007/s12630-014-0160-7. Epub 2014 Apr 17. PMID 24740312